CLINICAL TRIAL: NCT00260689
Title: A Randomized Study of Three Immunosuppressive Regimens in Treatment Naive Patients With Severe Aplastic Anemia: Horse ATG/CsA Taper vs Rabbit-ATG/CsA vs Alemtuzumab
Brief Title: Three Immunosuppressive Treatment Regimens for Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060034; 06-H-0034 (Other: NIH)
Record Dates: First submitted 2005-12-01; First posted 2005-12-01 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05-15

CONDITIONS: Immunosuppresion; Thrombocytopenia; Pancytopenia; Neutropenia
Keywords: Immunosuppression; T-cells; Hematopoiesis; Autoimmunity; Thrombocytopenia; Severe Aplastic Anemia; SAA
MeSH Terms: conditions — Thrombocytopenia; Pancytopenia; Neutropenia; Autoimmune Diseases; Anemia, Aplastic | interventions — Antilymphocyte Serum; Cyclosporine; Alemtuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Horse ATG/CsA taper (Experimental): h-ATG (Anti-thymocyte globulin (horse)) + 6 months CsA (Cyclosporine) followed by an 18 month CsA taper
  Interventions: Biological: Anti-thymocyte globulin (horse); Drug: Cyclosporine
- Rabbit ATG/CsA (Experimental): r-ATG (Anti-thymocyte globulin (rabbit)) + 6 months CsA (Cyclosporine)
  Interventions: Biological: Anti-thymocyte globulin (rabbit); Drug: Cyclosporine
- Alemtuzumab (Experimental): Alemtuzumab administered for 10 days
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Biological: Anti-thymocyte globulin (rabbit)
  Arms: Rabbit ATG/CsA
Biological: Anti-thymocyte globulin (horse)
  Arms: Horse ATG/CsA taper
Drug: Cyclosporine
  Arms: Horse ATG/CsA taper; Rabbit ATG/CsA
Drug: Alemtuzumab
  Other Names: Campath
  Arms: Alemtuzumab

SUMMARY:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and a hypocellular bone marrow. Allogeneic bone marrow transplantation offers the opportunity for cure in 70% of patients, but most patients are not suitable candidates for hematopoietic stem cell transplantation (HSCT) due to advanced age or lack of a histocompatible donor. For these patients, comparable long term survival is attainable with immunosuppressive treatment with anti-thymocyte globulin (ATG) and cyclosporine (CsA). However, of those patients treated with horse ATG(h-ATG)/CsA, one quarter to one third will not respond, and about 50% of responders relapse. Auto-reactive T cells may be resistant to the effect of ATG/CsA (non-responders), while in others residual auto-reactive T cells expand post-treatment, leading to hematopoietic stem cell destruction and recurrent pancytopenia (relapse). As long term survival is correlated to response rates and robustness of hematopoietic recovery, novel immunosuppressive regimens that can achieve hematologic response and decrease relapse rates are needed.

This trial will compare the effectiveness of three immunosuppressive regimens as first line therapies in patients with SAA with early hematologic response as the primary endpoint, as well as assess the role of extended CsA treatment after h-ATG in reducing numbers of late events of relapse and clonal evolution. Randomization is employed to obtain an equal distribution of subject to each arm; comparisons of early hematologic responses will be made among the rates observed among the three concurrent arms (rabbit-ATG [r-ATG] versus standard h-ATG; alemtuzumab vs standard h-ATG). For long course CSA, comparison of primary end points will be to well established historic relapse rate of 38% at 2-3 years and a cumulative rate of clonal evolution of 15%.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and a hypocellular bone marrow. Allogeneic bone marrow transplantation offers the opportunity for cure in 70% of patients, but most patients are not suitable candidates for hematopoietic stem cell transplantation (HSCT) due to advanced age or lack of a histocompatible donor. For these patients, comparable long term survival is attainable with immunosuppressive treatment with anti-thymocyte globulin (ATG) and cyclosporine (CsA). However, of those patients treated with horse ATG(h-ATG)/CsA, one quarter to one third will not respond, and about 50% of responders relapse. Auto-reactive T cells may be resistant to the effect of ATG/CsA (non-responders), while in others residual auto-reactive T cells expand post-treatment, leading to hematopoietic stem cell destruction and recurrent pancytopenia (relapse). As long term survival is correlated to response rates and robustness of hematopoietic recovery, novel immunosuppressive regimens that can achieve hematologic response and decrease relapse rates are needed.

This trial will compare the effectiveness of three immunosuppressive regimens as first line therapies in patients with SAA with early hematologic response as the primary endpoint, as well as assess the role of extended CsA treatment after h-ATG in reducing numbers of late events of relapse and clonal evolution. Randomization is employed to obtain an equal distribution of subject to each arm; comparisons of early hematologic responses will be made among the rates observed among the three concurrent arms (rabbit-ATG [r-ATG] versus standard h-ATG; alemtuzumab vs standard h-ATG). For long course CSA, comparison of primary end points will be to well established historic relapse rate of 38% at 2-3 years and a cumulative rate of clonal evolution of 15%.

In the original design subjects were randomized to one of three different regimens: h-ATG + 6 months CsA followed by an 18 month CsA taper; r-ATG + 6 months CsA; or alemtuzumab (Campath). Subjects failing to respond to r-ATG will be crossed over to alemtuzumab (Campath), and subjects failing alemtuzumab (Campath) will be crossed over to r-ATG. Subjects failing to respond to h-ATG + CsA taper will go off study and be evaluated for eligibility for a second course of immunosuppression on companion protocol 03-H-0249, which similarly randomizes subjects between r-ATG and alemtuzumab (Campath) as salvage therapy.

The Campath arm was closed to new accrual for lack of efficacy on 4/10/2008. Subsequently, new accruals will be randomized to h-ATG + 6 months CsA followed by an 18 month CsA taper or r-ATG + 6 months CsA. Subjects failing to respond to h-ATG + CsA taper will go off study and be evaluated for eligibility for a second course of immunosuppression on companion protocol 03-H-0249, which similarly randomizes subjects between r-ATG and alemtuzumab (Campath ) as salvage therapy. Subjects who fail to respond to r-ATG + 6 months CsA will be offered treatment with h-ATG as salvage therapy or will go off-study to alternative treatments or stem cell transplant (from sibling or unrelated donor).

The primary endpoint will be hematologic response, defined as no longer meeting criteria for SAA, at 6 months. Secondary endpoints are relapse, robustness of hematologic recovery at 6 months, response at 3 and 12 months, survival, clonal evolution to PNH, myelodysplasia and acute leukemia. Long-course CSA will be assessed separately for its efficacy in reducing late events of relapse and evolution by comparison to historical control data.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Severe aplastic anemia characterized by bone marrow cellularity less than 30% (excluding lymphocytes) and at least two of the following:

   * Absolute neutrophil count less than 500/microliter
   * Platelet count less than 20,000/microliter
   * Absolute reticulocyte count less than 60,000/microliter
2. Age greater than or equal to 2 years old
3. Weight greater than 12 kg

EXCLUSION CRITERIA:

1. Diagnosis of Fanconi's anemia
2. Evidence of a clonal disorder on cytogenetics. Patients with super severe neutropenia (ANC less than 200/microliter) will not be excluded initially if cytogenetics are not available or pending. If evidence of a clonal disorder is later identified, the patient will go off study.
3. Prior immunosuppressive therapy with ATG, ALG, alemtuzumab, or high dose cyclophosphamide.
4. Infection not adequately responding to appropriate therapy.
5. Serologic evidence of HIV infection.
6. Failure to discontinue the herbal supplements Echinacea purpurea or Usnea barbata (Old Man's Beard) within 2 weeks of enrollment.
7. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within 7-10 days is likely.
8. Potential subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible.
9. Current pregnancy, or unwillingness to take oral contraceptives or refrain from pregnancy if of childbearing potential.
10. Not able to understand the investigational nature of the study or give informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-11-28; Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Townsley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NIH Biomedical Translational Research Information System (BTRIS)

REFERENCES:
- [Background] Young NS, Barrett AJ. The treatment of severe acquired aplastic anemia. Blood. 1995 Jun 15;85(12):3367-77. No abstract available. PMID 7780125
- [Background] Young NS, Maciejewski J. The pathophysiology of acquired aplastic anemia. N Engl J Med. 1997 May 8;336(19):1365-72. doi: 10.1056/NEJM199705083361906. No abstract available. PMID 9134878
- [Background] Zoumbos NC, Gascon P, Djeu JY, Trost SR, Young NS. Circulating activated suppressor T lymphocytes in aplastic anemia. N Engl J Med. 1985 Jan 31;312(5):257-65. doi: 10.1056/NEJM198501313120501. PMID 2981406
- [Background] Feng X, Scheinberg P, Biancotto A, Rios O, Donaldson S, Wu C, Zheng H, Sato K, Townsley DM, McCoy JP, Young NS. In vivo effects of horse and rabbit antithymocyte globulin in patients with severe aplastic anemia. Haematologica. 2014 Sep;99(9):1433-40. doi: 10.3324/haematol.2014.106542. Epub 2014 Jun 6. PMID 24907357
- [Background] Scheinberg P, Townsley D, Dumitriu B, Scheinberg P, Weinstein B, Rios O, Wu CO, Young NS. Horse antithymocyte globulin as salvage therapy after rabbit antithymocyte globulin for severe aplastic anemia. Am J Hematol. 2014 May;89(5):467-9. doi: 10.1002/ajh.23669. Epub 2014 Mar 7. PMID 24415649
- [Background] Scheinberg P, Nunez O, Weinstein B, Scheinberg P, Wu CO, Young NS. Activity of alemtuzumab monotherapy in treatment-naive, relapsed, and refractory severe acquired aplastic anemia. Blood. 2012 Jan 12;119(2):345-54. doi: 10.1182/blood-2011-05-352328. Epub 2011 Nov 8. PMID 22067384
- [Background] Scheinberg P, Nunez O, Weinstein B, Scheinberg P, Biancotto A, Wu CO, Young NS. Horse versus rabbit antithymocyte globulin in acquired aplastic anemia. N Engl J Med. 2011 Aug 4;365(5):430-8. doi: 10.1056/NEJMoa1103975. PMID 21812672
- [Derived] Zaimoku Y, Patel BA, Adams SD, Shalhoub R, Groarke EM, Lee AAC, Kajigaya S, Feng X, Rios OJ, Eager H, Alemu L, Quinones Raffo D, Wu CO, Flegel WA, Young NS. HLA associations, somatic loss of HLA expression, and clinical outcomes in immune aplastic anemia. Blood. 2021 Dec 30;138(26):2799-2809. doi: 10.1182/blood.2021012895. PMID 34724566
- [Derived] Giudice V, Wu Z, Kajigaya S, Fernandez Ibanez MDP, Rios O, Cheung F, Ito S, Young NS. Circulating S100A8 and S100A9 protein levels in plasma of patients with acquired aplastic anemia and myelodysplastic syndromes. Cytokine. 2019 Jan;113:462-465. doi: 10.1016/j.cyto.2018.06.025. Epub 2018 Jun 27. PMID 29958797
- [Derived] Giudice V, Banaszak LG, Gutierrez-Rodrigues F, Kajigaya S, Panjwani R, Ibanez MDPF, Rios O, Bleck CK, Stempinski ES, Raffo DQ, Townsley DM, Young NS. Circulating exosomal microRNAs in acquired aplastic anemia and myelodysplastic syndromes. Haematologica. 2018 Jul;103(7):1150-1159. doi: 10.3324/haematol.2017.182824. Epub 2018 Apr 19. PMID 29674506
- [Derived] Hosokawa K, Kajigaya S, Feng X, Desierto MJ, Fernandez Ibanez MD, Rios O, Weinstein B, Scheinberg P, Townsley DM, Young NS. A plasma microRNA signature as a biomarker for acquired aplastic anemia. Haematologica. 2017 Jan;102(1):69-78. doi: 10.3324/haematol.2016.151076. Epub 2016 Sep 22. PMID 27658437
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0034.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Horse ATG/CsA Taper: Horse Anti-thymocyte Globulin (h-ATG) + 6 months Cyclosporine (CsA) followed by an 18 month CsA taper
- Rabbit ATG/CsA: Rabbit Anti-thymocyte Globulin (r-ATG) + 6 months Cyclosporine (CsA)
- Alemtuzumab: Alemtuzumab (Campath) administered for 10 days
Period: Overall Study
Arm/Group | Horse ATG/CsA Taper | Rabbit ATG/CsA | Alemtuzumab
Started | 60 | 60 | 16
Completed | 19 | 11 | 1
Not Completed | 41 | 49 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Horse ATG/CsA Taper | Rabbit ATG/CsA | Alemtuzumab | Total
Number analyzed (Participants) | 60 | 60 | 16 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 21 | 4 | 39
  Between 18 and 65 years | 38 | 35 | 8 | 81
  >=65 years | 8 | 4 | 4 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 4 | 54
  Male | 33 | 37 | 12 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 7 | 29
  Not Hispanic or Latino | 50 | 44 | 9 | 103
  Unknown or Not Reported | 1 | 3 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 20 | 1 | 36
  White | 29 | 24 | 7 | 60
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 9 | 14 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response
Description: Hematologic response is defined as subjects having blood counts no longer meeting the standard ("Camitta") criteria for severe pancytopenia in Severe Aplastic Anemia, equivalent to 2 of the following values obtained on 2 serial blood count measurements at least one week apart at landmark time points (3, 6 and 12 months)
  * Absolute neutrophil count > 500/ μL
  * Platelet count > 20,000/ μL
  * Reticulocyte count > 60,000/ μL
  Improvement in counts that are dependent upon exogenously administered growth factors or transfusion will not be considered as fulfilling response criteria.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Horse ATG/CsA Taper | Rabbit ATG/CsA | Alemtuzumab
Number analyzed (Participants) | 60 | 60 | 16
Participants | 38 | 20 | 3

2. Primary Outcome: Hematologic Response
Description: as for outcome 1
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Horse ATG/CsA Taper | Rabbit ATG/CsA | Alemtuzumab
Number analyzed (Participants) | 60 | 60 | 16
Participants | 41 | 22 | 3

3. Primary Outcome: Hematologic Response
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Horse ATG/CsA Taper | Rabbit ATG/CsA | Alemtuzumab
Number analyzed (Participants) | 60 | 60 | 16
Participants | 40 | 18 | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Horse ATG/CsA Taper | Rabbit ATG/CsA | Alemtuzumab
All-Cause Mortality (participants affected / at risk) | 11/60 | 18/60 | 7/16
Serious Adverse Events (participants affected / at risk) | 7/60 | 11/60 | 6/16
Other Adverse Events (participants affected / at risk) | 36/60 | 39/60 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Horse ATG/CsA Taper (N=60) | Rabbit ATG/CsA (N=60) | Alemtuzumab (N=16)
CNS hemorrhage/bleeding (Blood and lymphatic system disorders) | 0 | 1 | 0
Edema: limb (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac troponin I (Cardiac disorders) | 1 | 0 | 0
Hypertension (Cardiac disorders) | 0 | 1 | 0
Supraventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0
Serum sickness (Immune system disorders) | 2 | 4 | 0
Serum sickness/Infection (Immune system disorders) | 0 | 1 | 0
Infection (documented clinically or microbiologically with grade 3 or 4 neutropenia) (Infections and infestations) | 3 | 1 | 5
Infection without neutropenia (Infections and infestations) | 0 | 1 | 0
Creatinine (grade 2) (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Seizures (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Horse ATG/CsA Taper (N=60) | Rabbit ATG/CsA (N=60) | Alemtuzumab (N=16)
edema (Blood and lymphatic system disorders) | 0 | 1 | 0
edema - mild lower extremity (Blood and lymphatic system disorders) | 1 | 0 | 0
gingival hypertrophy (Blood and lymphatic system disorders) | 0 | 1 | 0
Hemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
lower extremity edema (Blood and lymphatic system disorders) | 0 | 1 | 0
lower extremity swelling (Blood and lymphatic system disorders) | 0 | 1 | 0
slight edema pitting (Blood and lymphatic system disorders) | 1 | 0 | 0
slight pitting edema (Blood and lymphatic system disorders) | 0 | 1 | 0
swelling (lower extremity) (Blood and lymphatic system disorders) | 1 | 0 | 0
swelling ankles (Blood and lymphatic system disorders) | 1 | 0 | 0
swelling feet and hands (Blood and lymphatic system disorders) | 0 | 1 | 0
bradycardia (Cardiac disorders) | 0 | 1 | 0
Edema, ankles (Cardiac disorders) | 2 | 1 | 0
Edema, lower legs (Cardiac disorders) | 3 | 1 | 1
fluid overload (Cardiac disorders) | 2 | 1 | 0
h Blood pressure (Cardiac disorders) | 1 | 0 | 0
h BP (Cardiac disorders) | 3 | 1 | 0
high blood pressure (Cardiac disorders) | 1 | 0 | 0
Hypertension (Cardiac disorders) | 8 | 9 | 3
hypotension (Cardiac disorders) | 2 | 3 | 0
i SBP (Cardiac disorders) | 1 | 0 | 0
irregular pulse (Cardiac disorders) | 0 | 1 | 0
S tachycardia (Cardiac disorders) | 0 | 1 | 0
substernal pressure (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1 | 1
Hot flashes (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism, subclinical (Endocrine disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
abdominal gas (Gastrointestinal disorders) | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
abdominal pain with loose stools (Gastrointestinal disorders) | 1 | 0 | 0
bleeding, swollen gums (Gastrointestinal disorders) | 0 | 1 | 0
bloated (Gastrointestinal disorders) | 1 | 0 | 0
decreased (Gastrointestinal disorders) | 0 | 1 | 0
dehydration (Gastrointestinal disorders) | 1 | 0 | 0
diarrhea (Gastrointestinal disorders) | 5 | 8 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 2 | 4 | 2
gingivial hyperplasia (Gastrointestinal disorders) | 0 | 1 | 0
gingivial hyperplasia - mild (Gastrointestinal disorders) | 1 | 0 | 0
gingivitis (Gastrointestinal disorders) | 0 | 1 | 0
gum hyperplasia (Gastrointestinal disorders) | 0 | 1 | 0
gum hypertrophy (Gastrointestinal disorders) | 0 | 1 | 0
Heartburn (Gastrointestinal disorders) | 3 | 1 | 1
i K+ (Gastrointestinal disorders) | 0 | 1 | 0
Indigestion (Gastrointestinal disorders) | 1 | 0 | 0
loose stool (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 0
nausea + vomiting (Gastrointestinal disorders) | 2 | 1 | 0
poor appetite (Gastrointestinal disorders) | 1 | 1 | 0
vomiting (Gastrointestinal disorders) | 2 | 3 | 0
Abdominal (General disorders) | 1 | 0 | 0
abdominal pain (General disorders) | 1 | 2 | 0
Abdominal, cramps (General disorders) | 0 | 1 | 0
body aches (General disorders) | 1 | 0 | 0
chest discomfort (General disorders) | 1 | 0 | 0
chest pain (General disorders) | 0 | 2 | 0
Chest pressure (General disorders) | 0 | 1 | 0
chest tightness (General disorders) | 1 | 0 | 0
chills (General disorders) | 0 | 1 | 0
chills/rigors (General disorders) | 0 | 1 | 0
epigastric pain (General disorders) | 0 | 1 | 0
fever (General disorders) | 6 | 5 | 0
Headache (General disorders) | 10 | 6 | 1
leg pain (General disorders) | 0 | 1 | 0
Localized, back (General disorders) | 0 | 1 | 0
Localized, feet (burning), knee (General disorders) | 0 | 1 | 0
Localized, low back (General disorders) | 1 | 0 | 0
Localized, soles of feet, legs (General disorders) | 1 | 0 | 0
Localized, Throat (General disorders) | 0 | 0 | 1
Localized, throat, abdomen (General disorders) | 0 | 0 | 1
Localized, Wrist, bilateral (General disorders) | 0 | 1 | 0
low back pain (General disorders) | 1 | 0 | 0
Myalgia (general) (General disorders) | 0 | 1 | 0
Myalgia, arthralgia (General disorders) | 0 | 1 | 0
Myalgia, back (General disorders) | 0 | 1 | 0
Myalgia, calves (General disorders) | 1 | 0 | 0
neutropenic fever (General disorders) | 2 | 3 | 0
retrosternal chest pain (General disorders) | 0 | 1 | 0
rigor (General disorders) | 1 | 0 | 0
rigors (General disorders) | 5 | 2 | 0
stomach discomfort (General disorders) | 0 | 1 | 0
tired (General disorders) | 0 | 1 | 0
weight gain (General disorders) | 2 | 2 | 0
weight increase (General disorders) | 1 | 0 | 0
weight loss (General disorders) | 0 | 1 | 0
Elevated LFT's (Hepatobiliary disorders) | 9 | 9 | 5
Elevated t. bili (Hepatobiliary disorders) | 5 | 6 | 0
flu-like symptoms (Immune system disorders) | 1 | 0 | 0
joint Pain (Immune system disorders) | 0 | 1 | 0
Labeled infusion related (Immune system disorders) | 28 | 31 | 15
Serum sickness (Immune system disorders) | 2 | 5 | 0
swelling (Immune system disorders) | 1 | 0 | 0
throat swelling (Immune system disorders) | 0 | 1 | 0
C. diff colitis (Infections and infestations) | 0 | 3 | 0
C. diff colitis and Blastocystis hominis (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 3 | 1 | 0
Mouth sores (Infections and infestations) | 3 | 3 | 1
Mouth sores (neg. Cxs) (Infections and infestations) | 0 | 1 | 0
Shingles (Infections and infestations) | 1 | 0 | 0
Trush (Infections and infestations) | 1 | 1 | 1
Upper Respiratory Tract (Infections and infestations) | 0 | 1 | 1
h ALT (Metabolism and nutrition disorders) | 1 | 1 | 0
h ALT/di bili (Metabolism and nutrition disorders) | 0 | 1 | 0
h AST (Metabolism and nutrition disorders) | 0 | 1 | 0
h creatinine (Metabolism and nutrition disorders) | 3 | 4 | 0
h creatinine -mild (Metabolism and nutrition disorders) | 1 | 0 | 0
h K (Metabolism and nutrition disorders) | 0 | 1 | 0
h LDH (Metabolism and nutrition disorders) | 0 | 1 | 0
h LFT (Metabolism and nutrition disorders) | 2 | 0 | 0
h LFT, creatinine (Metabolism and nutrition disorders) | 0 | 1 | 0
h LFTs (Metabolism and nutrition disorders) | 1 | 1 | 0
h PT, PTT (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglicemia (Metabolism and nutrition disorders) | 2 | 2 | 1
hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
hypertension (Metabolism and nutrition disorders) | 0 | 1 | 0
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
hypomagnesia (Metabolism and nutrition disorders) | 1 | 1 | 0
i magnesium (Metabolism and nutrition disorders) | 2 | 2 | 0
LFT abnormal (Metabolism and nutrition disorders) | 1 | 0 | 0
low albumin (Metabolism and nutrition disorders) | 0 | 1 | 0
renal failure (Metabolism and nutrition disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cramps (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
anxiety (Nervous system disorders) | 1 | 0 | 0
Anxiety, irritability (Nervous system disorders) | 0 | 1 | 0
dizziness (Nervous system disorders) | 0 | 1 | 0
Insomnia (Nervous system disorders) | 0 | 2 | 1
numbness (Nervous system disorders) | 1 | 0 | 0
Numbness fingers, wrists (Nervous system disorders) | 1 | 0 | 0
numbness/tingling (bilateral lower extremities) (Nervous system disorders) | 1 | 0 | 0
parastesias (Nervous system disorders) | 0 | 1 | 0
Perioral tingling (Nervous system disorders) | 1 | 0 | 0
Peripheral neuropathy, CsA induced (Nervous system disorders) | 0 | 1 | 0
tingling (Nervous system disorders) | 0 | 1 | 0
Tremor, hands (Nervous system disorders) | 0 | 1 | 0
tremors (Nervous system disorders) | 0 | 1 | 0
acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
mild renal insufficiency (Renal and urinary disorders) | 1 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
crackles (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
crackles in lungs (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
crackles lungs (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
dry cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
short of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
sob (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Body hair growth (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema, LE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
erythematous rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
hair growth (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
increased hair growth (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
itchy palms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
palm itching (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
palms slightly red (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
rash (arms) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
rash - mild (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
rash face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash, face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
rash, hives, itching (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
urticarial rash -mild (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Originally, there were 3 regimens: h-ATG/CsA ; r-ATG/CsA; alemtuzumab. Subjects not responding to r-ATG will cross over to alemtuzumab, and subjects failing alemtuzumab will cross over to r-ATG. Subjects not responding to h-ATG/CsA will go off study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes